CLINICAL TRIAL: NCT06775678
Title: A Single-centre Phase II Clinical Study of Spatially Fragmentation Radiotherapy Combined With Low-dose Radiotherapy for Reversal of Immunotherapy Combined With Chemotherapy Resistance in Locally Advanced Inoperable or Advanced Non-small Cell Lung Cancer
Brief Title: Spatial Fragmentation Combined With Low-dose Radiotherapy for Immunotherapy Combined With Chemotherapy-resistant Locally Advanced or Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20240009
Record Dates: First submitted 2025-01-08; First posted 2025-01-15 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancers; Radiation Treatment for Tumors
Keywords: Spatially Fractionated Radiation Treatment; low dose radiotherapy; Lung Cancers; Immunotherapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): 1. Patients received dose-specific irradiation using a medical linear accelerator to create each sphere of approximately 0.5 to 1.5 cm in diameter within the gross tumour volume (GTV) of the largest tumour, with spheres spaced 2.0 to 5.0 cm apart from each other as the high-dose area; the rest of the GTV was used as the low-dose area.
     For a single lesion, spatially divided radiotherapy was given, with the prescribed dose for the high-dose area: 800-1200cGy×3f, and the prescribed dose for the low-dose area: 100-300cGy×5f; all the remaining irradiable metastatic foci were given low-dose radiotherapy (palliative radiotherapy was given to the brain and bone metastases in accordance with the clinical routine, and was excluded from the scope of low-dose radiotherapy), with the prescribed dos
  2. During or within 1 week after radiotherapy, chemotherapy combined with immunotherapy was carried out according to the physical, pathological and genetic detection of the patients.
  Interventions: Radiation: Spatially Fractionated Radiation Therapy Combined With Low-dose Radiotherapy
- control group (Active Comparator): The control group only received conventional radiotherapy for chest or other lesions, followed by immunotherapy and chemotherapy according to the tumor stage, tolerance and genetic characteristics of the patients
  Interventions: Radiation: Conventional fractionated radiotherapy

INTERVENTIONS:
Radiation: Spatially Fractionated Radiation Therapy Combined With Low-dose Radiotherapy — Spatially Fractionated Radiation Therapy Combined With Low-dose Radiotherapy
  Arms: experimental group
Radiation: Conventional fractionated radiotherapy — Conventional fractionated radiotherapy
  Arms: control group

SUMMARY:
The purpose of this study was to evaluate the effect of immunotherapy combined with spatial fractionation radiotherapy and low dose radiotherapy on the prognosis of patients with advanced lung cancer under specific dose regimens (spatial fractionation radiotherapy: high dose region: 800-1200cGy × 3f, low dose region: 100-300cGy × 5f; low dose radiotherapy area: 100-300cGy × 5f). Through the phase II clinical trial, to determine the efficacy and safety of the combined treatment model in advanced lung cancer and its effect on the immune microenvironment of patients, so as to provide scientific basis for the optimization of treatment regimen for advanced lung cancer.

DETAILED DESCRIPTION:
The eligible subjects were randomly divided into the experimental group and the control group according to the proportion of 1:1. The experimental group was treated with space fractionation radiotherapy for a single lesion, with a prescription dose of 800-1200cGy × 3f in the high-dose area and 100-300cGy × 5f in the low-dose area. All other irradiable metastatic foci were given low-dose radiotherapy (brain and bone metastases were given palliative radiotherapy according to clinical routine, but not within the range of low-dose radiotherapy). The prescription dose was 100-300cGy × 5f. Chemotherapy combined with immunotherapy was given during or within 1 week after radiotherapy. The control group only received conventional radiotherapy for chest or other lesions, followed by immunotherapy and chemotherapy according to the tumor stage, tolerance and genetic characteristics of the patients. Peripheral blood routine, immune cell (lymphocyte) subsets and related cytokines were detected before radiotherapy, on the day after radiotherapy and within 7 days after 1 cycle of immunotherapy. Before radiotherapy and after 1 cycle of immunotherapy, the metastatic focus was biopsied, fixed with 4% formaldehyde for 12-24 hours, dehydrated by gradient alcohol in the dehydrator, and finally embedded in paraffin to make wax blocks for preservation. The toxic and side effects of the treatment were recorded in detail, and the symptomatic treatment and detailed records can be made according to the severity. Patients with severe adverse reactions (SAE) will stop treatment and report to the research center for inclusion in the statistics. The toxicity and side effects were evaluated by CTCAE5.0 standard, and the long-term side effects were evaluated by RTOG long-term toxicity evaluation criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form.
2. Be at least 18 years old.
3. Have a Karnofsky Performance Status (KPS) score of 70 or higher and an expected survival of more than 3 months.
4. Have histopathological evidence of small cell lung cancer, lung adenocarcinoma, or lung squamous cell carcinoma.
5. Have received prior immunotherapy and experienced disease progression.
6. The site targeted for radiotherapy has not been previously irradiated or it has been at least 6 months since the last radiotherapy.

Exclusion Criteria:

1. The patient has lesions that are not suitable for radiotherapy: malignant pleural effusion, ascites, meningeal metastasis, etc.
2. The patient has other serious comorbidities, such as myocardial infarction occurring within 6 months, severe arrhythmia, mental illness, etc., is unable to complete the treatment, or has an expected survival period of less than 3 months.
3. The patient has severe organ dysfunction, such as liver failure, cardiopulmonary failure, etc., and is difficult to tolerate radiotherapy.
4. The patient currently has a severe infection.
5. The patient has a known or suspected active autoimmune disease (congenital or acquired), such as uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, thyroiditis, etc. (Patients with vitiligo or those with cured childhood asthma can be included; patients with type 1 diabetes who have good insulin control can also be included).
6. The patient has experienced grade 3 or above cardiac or liver toxicity reactions or grade 4 toxicity reactions in other organs during previous immunotherapy.
7. Other situations where reviewers consider there are sufficient reasons for disqualification from the registered study: such as potential situations inconsistent with the clinical protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2028-01-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From enrollment to the end of treatment at 6 mouths

SECONDARY OUTCOMES:
Disease control rate | From enrollment to the end of treatment at 6 mouths
Progression free survival | From enrollment to the end of treatment at 6 mouths
Overall survival | From enrollment to the end of treatment at 6 mouths
Adverse Event | From enrollment to the end of treatment at 6 mouths

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided